CLINICAL TRIAL: NCT05184868
Title: Phase 1 Randomized, Double-blind, Three Period, Crossover Study Comparing PD/PK, Safety and Tolerability Profiles for Arecor Ultra-rapid Insulin Aspart (AT247), NovoLog® and Fiasp® in Participants With T1DM During CSII
Brief Title: AT247, NovoLog® and Fiasp® Administered Via Continuous Subcutaneous Infusion in Glucose Clamp Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arecor Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARE-247-103
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AT247 (Experimental): 0.02 U/Kg/H Basal via continuous subcutaneous infusion with 2 bolus 0.15 U/Kg doses in a glucose clamp for one 3-day period
  Interventions: Drug: AT247; Drug: NovoLog; Drug: Fiasp
- NovoLog® (Active Comparator): 0.02 U/Kg/H Basal via continuous subcutaneous infusion with 2 bolus 0.15 U/Kg doses in a glucose clamp for one 3-day period
  Interventions: Drug: AT247; Drug: NovoLog; Drug: Fiasp
- Fiasp® (Active Comparator): 0.02 U/Kg/H Basal via continuous subcutaneous infusion with 2 bolus 0.15 U/Kg doses in a glucose clamp for one 3-day period
  Interventions: Drug: AT247; Drug: NovoLog; Drug: Fiasp

INTERVENTIONS:
Drug: AT247 — Ultra rapid acting prandial insulin aspart
Drug: NovoLog — Rapid acting prandial insulin aspart
  Other Names: NovoRapid
Drug: Fiasp — Fast acting prandial insulin aspart

SUMMARY:
Phase 1 randomized, double-blind, three period, crossover study comparing the pharmacodynamic, pharmacokinetic, safety and tolerability profiles for Arecor ultra-rapid insulin aspart (AT247), NovoLog® and Fiasp® in participants with type 1 diabetes mellitus (T1DM) during continuous subcutaneous infusion (CSII)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with T1DM for at least 12 months.
2. Subjects who have been using an approved insulin pump or use multiple daily injections with basal and bolus insulin, with a stable total insulin dose <1.2 U/kg/day and bolus insulin dose <0.7 U/kg/day for at least 3 months.
3. Fasting C-peptide concentration of ≤0.3 nmol/l (0.9061 ng/ml), assessed at a plasma glucose concentration >90 mg/dL.
4. HbA1c concentration of ≤8.5% (≤69 mmol/mol).
5. BMI within the range ≥18.5 - ≤28.0 kg/m2.

Exclusion Criteria:

1. Known or suspected hypersensitivity to IMP or related products.
2. History or presence of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any in-situ carcinomas are allowed.
3. Clinically significant concomitant disease including cardiovascular, renal, hepatic, respiratory, gastrointestinal, hematological, dermatological, neurological, psychiatric, systemic or infections disease as judged by the investigator.
4. Supine blood pressure at screening (after resting for at least 5 min in supine position) outside the ranges for systolic 95-140 mmHg blood pressure and/or for diastolic blood pressure greater than 90 mmHg.
5. Smoking more than 5 cigarettes per day or equivalent use of any tobacco containing product, and unable to refrain from smoking during the in-house periods of the study. A positive urine cotinine test at screening and check-in.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Area under Curve for serum insulin | 0-30 minutes
Area under Curve for Glucose Infusion Rate | 0-60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento, Inc, Chula Vista, California, United States